CLINICAL TRIAL: NCT06179914
Title: Validation of Resilience Models About Cancer in Adolescence and Youth in Taiwan
Brief Title: Resilience Models in Adolescence and Youth With Cancer in Taiwan
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-SV(I)-20200060
Record Dates: First submitted 2023-11-23; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-11

CONDITIONS: Childhood Cancer; Coping Behavior; Hope; Resilience
Keywords: Resilience; Hope; social support; Coping; adolescent and young adult; uncertainty
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescence and Youth with cancer: Participants were diagnosed with cancer before 18 years old and aged between 10 and 24 years

SUMMARY:
Validation of Resilience Models about Cancer in Adolescence and Youth in Taiwan

DETAILED DESCRIPTION:
This study uses the disease resilience model as a framework to explore the relationship between physical, mental, spiritual, and social aspects of resilience in adolescents with cancer and to verify the resilience model. It is expected that the research results will serve as a reference for designing nursing interventions in the future and develop local Resilience model to improve quality of care.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with cancer before 18 years old
* Aged between 10 and 24 years
* Received cancer treatment or completed treatment

Exclusion Criteria:

* Diagnosis of mental problems (developmental delay or psychiatric illness)
* At the end of life

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: childhood cancer at age between 10 and 24
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Herth Hope Index (HHI) | 1 year
  Herth Hope Index (HHI) has 12 items. The12 items developed by Herth (1992) measures adults hope and contains three factors: cognitive-temporal (positive and desired outcome in the future), affective-behavioral (a feeling of confident with the reality-based goals and desirable outcomes), and affiliative-contextual (interconnect between self and others)(Herth, 1992). A higher score indicates a higher degree of hope.
Resilience in Illness Scale (HARS) | 1 year
  HARS is a single factor scale, consisting of 13 items that measure how participants feel or think about managing their health since diagnosis. The internal consistency reliability (0.84 to 0.86) and content validity have been tested by previous qualitative research (Haase & Marcia, 1994; Haase & Philips, 2004). Participants are asked to mark how much they agree or disagree with each sentence using response options from 1 (strongly disagree) to 6 (strongly agree) (Haase, et al., 1999). Higher total scores indicate a higher degree of resilience.

SECONDARY OUTCOMES:
Symptom Distress Scale (SDS) | 1 year
  SDS is developed from McCorkle & Young (1978), with a total of 13 questions, using a 1-5 scoring method. Higher of the total score, the higher the degree of symptom distress. The reliability of the instrument (r=.79-.89), using Ware's health perception scale test (r=0.9) (McCorkle, 1978). The reliability of the revised Chinese version is (Cronbach's α =.91-.96), the content validity index (CVI) is 0.95, and the readability is 0.95 (Lai, 1998). Higher total scores indicate a higher degree of symptom distress.
mishel Uncertainty in Illness Scale - Revised | 1 year
  It is developed from the uncertainty scale developed by Mishel, 1981, with a total of 33 questions. The reliability of the instrument is 0.91. The reliability of each scale ranges from 0.64-0.89, and its validity has been verified through theory (Mishel, 1981). The internal consistency reliability of the Chinese version of the literature is Cronbach's α =0.87, the internal consistency of the subscales is 0.85 and 0.66, and the simultaneous validity is 0.571 (Xu & Huang, 1996). Higher total scores indicate a higher degree of uncertainty.
Jalowiec Coping Scale-Revised | 1 year
  It is developed from Jalowiec et al, (1984). There are 40 items. The test-retest reliability of the instrument is 0.79. The internal consistency within the subscale is between 0.85-0.86. The total scale α=0.78 and the subscale is 0.84 (question solution), 0.83 (defensive behavior) (Jalowiec et al, 1984).Higher total scores indicate a higher frequency of used coping behaviors.
Spiritual Perspective Scale (SPS) | 1 year
  The SPS was developed from Jalowiec et al, (1984). There are 40 questions in total. The test-retest reliability of the instrument is 0.79. The internal consistency within the subscale is between 0.85-0.86. The total scale α=0.78 and the subscale is 0.84 (question solution), 0.83 (defensive behavior) (Jalowiec et al, 1984).
Perceived Social Support (PSS) | 1 year
  It is developed from the Perceived Family Support Scale of Procidano & Heller (1983). The scale has 20 questions and Cronbach's alpha reliability coefficients are .88 and 0.91 (Procidano & Heller, 1983; Puskar & Bernardo, Stark, 2008).Higher total scores indicate a higher social support.
Family Strengths | 1 year
  It is developed by Olson, McCubbin, Barnes, Larsen, Muxen, & Wilson (1985). There are 12 questions in the scale, and the items are: family self-esteem, family trust, family loyalty, family problem-solving ability, question options range from strongly agree to strongly disagree, the score range is from 12 to 60, the higher the score, the higher the family strength, the alpha reliability coefficients are .73 and .88, Test-retest reliability was .73 and .79.
Self-Transcendence Scale | 1 year
  There are 15 questions, scored from 1 to 4. The higher the score, the higher the self-transcendence ability. The Cronbach's alpha reliability coefficient of the tool is .70-.94 (Chen, 2009); the pretest Cronbach's alpha reliability coefficient of the Chinese version of the literature is. 79, and the post-test Cronbach's alpha reliability coefficient is .78 (Chen, 2009).
Family Adaptability and Cohesion Scale | 1 year
  It is developed from Olson, et al, (1985), with a total of 30 questions. The reliability of the instrument is .87 (cohesion) and .78 (adaptability) (Olson et al, 1985); the Chinese version of the document Cronbach's α>0.6 (Fei, 1991).The higher the score is, the higher the family adaptability and cohesionself-transcendence.
Parent-Adolescent Communication | 1 year
  It is developed from Olson, McCubbin, Barnes, Larsen, Muxen, & Wilson, (1985). There are 30 questions, which can be divided into two subscales, with reliabilities of 0.87 and 0.78 respectively, using the confirmatory factor analysis (Olson et al. ,1985). The Cronbach's alpha coefficient of the Chinese version of the father-child communication questionnaire is .76, the Cronbach's alpha coefficient of the mother-child communication questionnaire is .84(Chen, 2001). Higher scores indicate better communication.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yu J, Dong H, Song Y, Zhu F. Influencing Factors of Hope Among Chinese Patients With Hematological Malignancies From the Perspective of Positive Psychology: A Cross-sectional Study. Cancer Nurs. 2022 Nov-Dec 01;45(6):465-472. doi: 10.1097/NCC.0000000000001035. Epub 2022 Jan 13. PMID 35025774
- [Result] Yu J, Song H. Prevalence and risk factors of loneliness among patients with hematological malignancies. Medicine (Baltimore). 2022 Dec 2;101(48):e31900. doi: 10.1097/MD.0000000000031900. PMID 36482642
- [Result] Borrescio-Higa F, Valdes N. The Psychosocial Burden of Families with Childhood Blood Cancer. Int J Environ Res Public Health. 2022 Jan 5;19(1):599. doi: 10.3390/ijerph19010599. PMID 35010854
- [Result] Linder LA, Hooke MC. Symptoms in Children Receiving Treatment for Cancer-Part II: Pain, Sadness, and Symptom Clusters. J Pediatr Oncol Nurs. 2019 Jul/Aug;36(4):262-279. doi: 10.1177/1043454219849578. PMID 31307323
- [Result] Sharp K, Tillery R, Long A, Wang F, Pan H, Phipps S. Trajectories of resilience and posttraumatic stress in childhood cancer: Consistency of child and parent outcomes. Health Psychol. 2022 Apr;41(4):256-267. doi: 10.1037/hea0001132. Epub 2021 Dec 2. PMID 34855418
- [Result] Rosales P, Evangelista L, Guo Y, Agbayani CG, Kain ZN, Fortier MA. Exploring Differences in Perceived Satisfaction, Resilience, and Achievement Between Hispanic and Non-Hispanic White Childhood Cancer Survivors. J Pediatr Health Care. 2021 Mar-Apr;35(2):196-204. doi: 10.1016/j.pedhc.2020.10.003. Epub 2021 Jan 28. PMID 33516620
- [Result] Li Y, Ni N, Zhou Z, Dong J, Fu Y, Li J, Luan Z, Peng X. Hope and symptom burden of women with breast cancer undergoing chemotherapy: A cross-sectional study. J Clin Nurs. 2021 Aug;30(15-16):2293-2300. doi: 10.1111/jocn.15759. Epub 2021 Mar 23. PMID 33756013
- [Result] Taylor EJ, Petersen C, Oyedele O, Haase J. Spirituality and Spiritual Care of Adolescents and Young Adults with Cancer. Semin Oncol Nurs. 2015 Aug;31(3):227-41. doi: 10.1016/j.soncn.2015.06.002. Epub 2015 Jun 6. PMID 26210201
- [Result] Haase JE. The adolescent resilience model as a guide to interventions. J Pediatr Oncol Nurs. 2004 Sep-Oct;21(5):289-99; discussion 300-4. doi: 10.1177/1043454204267922. PMID 15381798
- [Result] Decker C, Phillips CR, Haase JE. Information needs of adolescents with cancer. J Pediatr Oncol Nurs. 2004 Nov-Dec;21(6):327-34. doi: 10.1177/1043454204269606. PMID 15475469
- [Result] Laksmita OD, Chung MH, Liao YM, Haase JE, Chang PC. Predictors of resilience among adolescent disaster survivors: A path analysis. J Adv Nurs. 2020 Aug;76(8):2060-2071. doi: 10.1111/jan.14396. Epub 2020 May 19. PMID 32301129